CLINICAL TRIAL: NCT04553120
Title: Improving the Exposure Therapy Through Projection-based Augmented Reality for the Treatment of Cockroach Phobia: A Multiple-baseline Single Case Study
Brief Title: Improving the Exposure Therapy Through Projection-based Augmented Reality for the Treatment of Cockroach Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N1256
Record Dates: First submitted 2020-07-01; First posted 2020-09-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Animal Phobia
Keywords: Specific Phobia; Cockroach phobia; Exposure therapy; Augmented Reality; Projection-Based; Single case study
MeSH Terms: conditions — Zoophobia; Phobia, Specific

STUDY DESIGN:
Intervention Model Description: Single case, multiple-baseline AB design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alternating treatments condition - 10 days wait (Experimental): The intervention will be based on exposure therapy to cockroaches using P-ARET. Main components: Psychoeducation, Exposure to the feared object (cockroach), modeling (the therapist will interact with the phobic stimulus first and if possible, the patient will follow the same steps), cognitive restructuring, and reinforcement and relapse prevention.
  Interventions: Behavioral: Alternating single stimulus and multiple stimuli
- Alternating treatments condition - 9 days wait (Experimental): The intervention will be based on exposure therapy to cockroaches using P-ARET. Main components: Psychoeducation, Exposure to the feared object (cockroach), modeling (the therapist will interact with the phobic stimulus first and if possible, the patient will follow the same steps), cognitive restructuring, and reinforcement and relapse prevention.
  Interventions: Behavioral: Alternating single stimulus and multiple stimuli
- Alternating treatments condition - 13 days wait (Experimental): The intervention will be based on exposure therapy to cockroaches using P-ARET. Main components: Psychoeducation, Exposure to the feared object (cockroach), modeling (the therapist will interact with the phobic stimulus first and if possible, the patient will follow the same steps), cognitive restructuring, and reinforcement and relapse prevention.
  Interventions: Behavioral: Alternating single stimulus and multiple stimuli
- Alternating treatments condition - 12 days wait (Experimental): The intervention will be based on exposure therapy to cockroaches using P-ARET. Main components: Psychoeducation, Exposure to the feared object (cockroach), modeling (the therapist will interact with the phobic stimulus first and if possible, the patient will follow the same steps), cognitive restructuring, and reinforcement and relapse prevention.
  Interventions: Behavioral: Alternating single stimulus and multiple stimuli

INTERVENTIONS:
Behavioral: Alternating single stimulus and multiple stimuli — P-ARET for cockroach phobia alternating between two interventions: exposure to a single stimulus (always using the same projected cockroach) and exposure to multiple stimuli (different cockroaches in terms of number, shape, colour and movement). It will be counterbalanced to start the same number of participants in each of the two modalities. The two conditions will be randomly applied for each participant, with the restriction of that each condition will be applied 3 times.
  There will be 6 weekly sessions of approximately 1 hour. The purpose of this exposure treatment is to confront patients to the phobic stimuli in a controlled manner, which favors the habituation process and allows them to accept that the negative consequences they fear do not actually occur. All exposure sessions should be recorded (patients will sign informed consent for recording prior to treatment initiation).

SUMMARY:
The aim of this study is to test the efficacy and efficiency of varying the phobic stimuli during the augmented reality (AR) exposure therapy using multiple stimuli versus one single stimulus through projection-based AR (P-ARET) for the treatment of participants diagnosed with cockroach phobia.

DETAILED DESCRIPTION:
Specific phobia (SP) refers to an extreme and persistent fear of a specific object or situation that is out of proportion to the actual danger or threat. SP is the most prevalent anxiety disorder with substantial impairment and comorbidity. Animal fear is one of the most prevalent subtypes of SP. In vivo exposure is the treatment of choice for this problem, but this technique is associated to limitations in its implementation related to the access and acceptability (i.e., low acceptance on the part of patients and therapists, high dropout rates, limited access to the treatment and, difficulties in its application in the clinical context). Augmented Reality (AR) offers some advantages in delivering the exposure technique: 1) Exposure to multiple virtual stimuli; 2) Going beyond reality; 3) Allowing complete control over the situation; 4) It allows privacy and confidentiality. Particularly, the most significant aspect of AR is that the virtual elements add relevant and helpful information to the physical information available in the real world.

The study will follow the guidelines of a multiple-baseline single case design with alternating treatments. Participants (N = 4) who received a diagnosis of SP for cockroaches (DSM-5), will be randomly assigned to different baselines (ranging between 8 and 14 days) and all of them will receive the two experimental conditions: 1) AR exposure therapy with multiple stimuli and; 2) AR exposure therapy with a single stimulus. Five evaluation moments will be included: pre-intervention (baseline), post- intervention, and follow-up at the first month, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Meeting DSM-5 diagnostic criteria for SP (animal subtype) to cockroaches
* Having a minimum of six-month duration of the phobia
* Sign an informed consent
* Presenting a score of at least 4 on the fear and avoidance scales of the diagnostic interview applied

Exclusion Criteria:

* Presence of another severe mental disorder that requires immediate attention
* Having current alcohol or drug dependence or abuse, psychosis or severe organic illness
* Currently being treated in a similar treatment program
* Being capable of inserting their hands in a plastic container with a cockroach (during the behavioral test)
* Receiving other psychological treatment during the study for cockroach phobia
* Start receiving pharmacological treatment during the study (or in case of being already taking them, change the drug or dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Avoidance Test (BAT; adapted from Öst, Salkovskis, & Hellström's, 1991) | At the beginning of the intervention and immediately after the treatment
  Patients will be confronted to a real cockroach and they will be encouraged to get closer and interact with the stimulus as much as they can. The anxiety level (0-10), distance and level of interaction with the animal will be registered evaluated in a scale ranging from 0 (the participant does not enter the room) to 12 (interacts with the cockroach).
Change in fear, avoidance, belief in negative thoughts and coping ability with the feared stimulus levels. | Once a day (from the start of the baseline until the end of the treatment) and at 1, 6 and 12 months after the end of the treatment.
  Item1: If you see a cockroach in front of you at this moment… To what extent would you be scared of it? Item 2: If you see a cockroach in front of you at this moment… to what extent would you avoid it?, Item 3: If you see a cockroach in front of you at this moment… To what extent would you believe that it is dangerous for you?, Item 4: To what extent you believe that you could cope with a cockroach of different size, colour and shape? Ranged from 0 (nothing) to 10 (very much)

SECONDARY OUTCOMES:
Change in Fear of Cockroaches Questionnaire (adapted from Fear of Spiders Questionnaire; FSQ, Szymanski & O'Donohue, 1995) | At the beginning of the intervention and immediately after the treatment
  This questionnaire assesses the level of fear to cockroaches. It has 18 items evaluated in a scale ranging from 1 (nothing) to 7 (very much).
Patient's Improvement Scale (adapted from the Clinical Global Impression scale; CGI, Guy, 1976). | At the beginning of the intervention and immediately after the treatment
  This instrument evaluates the degree of improvement of the patient' symptoms after the treatment compared to the start. It is ranged from 1 (much worse) and 7 (much better).
Change in Behavioral Avoidance Test through AR (BAT; adapted from Öst, Salkovskis, & Hellström's, 1991) | At the beginning of the intervention and immediately after the treatment
  Patients will be confronted to a novel projected cockroach (not used before in any treatment condition) and they will be encouraged to get closer and interact with the stimulus as much as they can. The anxiety level (0-10), distance and level of interaction with the animal will be registered evaluated in a scale ranging from 0 (the participant does not enter the room) to 12 (interacts with the cockroach).
Preferences | Immediately after the treatment
  Preferences about the treatment condition (MS versus SS) were assessed with a questionnaire composed of the following items: Item 1 "If you could choose between the two types of exposure sessions, which one would you choose?; Item 2 "Which of these two ways of applying the exposure session do you consider to be more effective in helping you overcome your problem?"; Item 3 "Which of these two ways of applying the exposure session do you consider more aversive?"; and Item 4 "Which of these two ways to apply the exposure session would you recommend to a friend who had the same problem?"

OTHER OUTCOMES:
Change in Anxiety Disorders Interview Schedule for DSM-IV-TR (ADIS-IV) - Specific Phobia | At the beginning of the intervention and immediately after the treatment, and at 1, 6 and 12 months after the end of the treatment.
  Diagnostic interview for specific phobia based on DSM-IV-TR criteria.
Change in The Clinician Severity Scale (adapted from Di Nardo, Brown & Barlow, 1994). | At the beginning of the intervention and immediately after the treatment
  This instrument assesses the severity of symptoms evaluated by the clinician and the scale ranged from 0 (absent) to 8 (very severe).
Change in Scale of expectation and satisfaction with the treatment (adapted from Borkovec y Nau, 1972) | At the beginning of the intervention and immediately after the treatment
  This instrument contains 6 items ranged from 0 (nothing) to 10 (very much) assessing the patient's opinions about the treatment, focusing on their expectations and degree of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shiban Y, Schelhorn I, Pauli P, Muhlberger A. Effect of combined multiple contexts and multiple stimuli exposure in spider phobia: A randomized clinical trial in virtual reality. Behav Res Ther. 2015 Aug;71:45-53. doi: 10.1016/j.brat.2015.05.014. Epub 2015 May 28. PMID 26072451
- [Background] Wrzesien, M., Botella, C., Bretón-López, J., del Río González, E., Burkhardt, J. M., Alcañiz, M., & Pérez-Ara, M. Á. (2015). Treating small animal phobias using a projective-augmented reality system: A single-case study. Computers in Human Behavior, 49, 343-353.
- [Background] Botella C, Mira A, Moragrega I, Garcia-Palacios A, Breton-Lopez J, Castilla D, Riera Lopez Del Amo A, Soler C, Molinari G, Quero S, Guillen-Botella V, Miralles I, Nebot S, Serrano B, Majoe D, Alcaniz M, Banos RM. An Internet-based program for depression using activity and physiological sensors: efficacy, expectations, satisfaction, and ease of use. Neuropsychiatr Dis Treat. 2016 Feb 23;12:393-406. doi: 10.2147/NDT.S93315. eCollection 2016. PMID 27042067